CLINICAL TRIAL: NCT06494904
Title: ED-Initiated Standard Versus High Dose Buprenorphine Induction
Brief Title: Standard Versus High Dose ED-Initiated Buprenorphine Induction
Acronym: ED-ENVISION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Drug Abuse Treatment Clinical Trials Network (Network); The Emmes Company, LLC (Industry); National Institute on Drug Abuse (NIDA) (NIH); Alameda Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UG1DA015831 (NIH); UG1DA015831 (NIH)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder
Keywords: Buprenorphine; Substance use disorder treatment
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is a multi-site double-blind, double-dummy randomized clinical trial. Only the DSC staff overseeing the random assignment schedule, a few designated CCC staff, and the central research staff preparing the study medication will be unblinded; all other study personnel and participants will remain blinded to treatment arm until the nationwide completion of the trial and the database is formally locked. Detailed information on the study procedures regarding the double-blinding will be contained in a standalone Blinding Management Plan and Study Site Blinding Plan. A DSMB will review study data throughout the course of the trial in a blinded fashion (e.g., masked treatment assignments), however they can request to be unblinded at any time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose SL-BUP (Experimental): Participants will receive three 5.7 mg Zubsolv pills; all will be active medication.
  Interventions: Drug: Buprenorphine
- Standard SL-BUP (Active Comparator): Participants will receive three pills; one 5.7 mg Zubsolv pill with active medication and two placebo pills.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — All patients will receive 3 pills and will be observed for 2 hours post-study medication administration with repeated COWS at approximately hours 1 and 2. All participants will be given a referral for ongoing MOUD and will be discharged with a prescription for 16 mg daily of buprenorphine daily.
  Other Names: Zubsolv

SUMMARY:
This study is a multisite double-blind, double-dummy, randomized clinical trial enrolling ED patients with untreated moderate to severe opioid use disorder (OUD) to compare Standard Dose Induction (SDI) and High Dose Induction (HDI) on rates of participation in OUD treatment within 10 days post randomization, and opioid withdrawal symptoms, opioid craving, and use of illicit and non-prescribed drugs.

DETAILED DESCRIPTION:
This study will recruit, train, and provide resources to approximately 4 ED systems throughout the U.S. to recruit ED patients presenting with OUD not receiving medications for opioid use disorder (MOUD) as part of an RCT to compare SDI (Zubsolv 5.7/1.4 mg buprenorphine/naloxone* plus 2 placebo tablets) with HDI (three Zubsolv 5.7/1.4 mg* buprenorphine/naloxone tablets) to evaluate rate of participation in OUD treatment within 10 days post-randomization and differences in outcomes of tolerability, opioid withdrawal symptoms, craving, and use of illicit drugs.

ELIGIBILITY:
Inclusion Criteria:

All patients enrolled into the study must:

1. Be 18-65 years of age.
2. Be treated in the ED during study screening hours.
3. Meet DSM-5 diagnostic criteria for moderate to severe OUD.
4. Have a Clinical Opiate Withdrawal Scale (COWS) score of ≥8 at enrollment (including 2 objective signs of withdrawal at enrollment).
5. Have a urine toxicology test that is positive for opioids.
6. Be able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

All patients enrolled into the study must not:

1. Have a medical or psychiatric condition that requires hospitalization at the time of index ED visit.
2. Have a known hypersensitivity reaction to buprenorphine/naloxone
3. Be actively suicidal or severely cognitively impaired precluding informed consent.
4. Require ongoing prescription for opioid analgesics.
5. Have a physical exam or reported history consistent with severe liver failure
6. Have a positive urine test for methadone and reported use in the past 72 hours
7. Be a prisoner or in police custody at the time of index ED visit.
8. Be unwilling to follow study procedures (e.g., unwilling to provide permission to contact referral provider/program or unavailable for the follow-up assessments)
9. Have prior enrollment in the current study.
10. Receiving MOUD treatment within the past 7 days.
11. Be pregnant as determined by human gonadotropin (hCG) testing at the index ED visit
12. Have a respiratory rate <8 or oxygen saturation <93%
13. Be a participant in any other clinical trial in which medications are being delivered or the use of an investigational drug or device within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Engagement in Treatment (10) | Within 10 days after study randomization
  The proportion of patients in each of the two study arms participating in OUD treatment within 10 days after the study randomization

SECONDARY OUTCOMES:
Craving | Measured daily for 10 days post randomization
  The maximum intensity of opioid cravings during the preceding 24 hours assessed daily for 10 days post randomization using a numerical rating scale (0 to 10).
Withdrawal | Measured daily for 10 days post randomization
  The maximum intensity of opioid withdrawal symptoms during the preceding 24 hours assessed daily for 10 days post randomization using a numerical rating scale (0 to 10).
Substance Use | Measured daily for 10 days post randomization
  The number of days with illicit opioid and other substance use based on self-reported data obtained daily during the first 10 days post randomization
Engagement in Treatment (30) | Within 30 days after randomization
  The proportion of patients in each of the two study arms participating in OUD treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gail D'Onofrio, MD, MS, Principal Investigator — Yale University; Kathryn Hawk, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - Highland Hospital, Oakland, California
  - San Leandro Hospital, San Leandro, California
  - Maine Medical Center, Portland, Maine
  - Cooper University Hospital, Camden, New Jersey
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
In line with the National Institutes of Health Helping to End Addiction Long-term (NIH HEAL) Initiative Public Access and Data Sharing Policy, publications and underlying primary data will be made available to the public.
Time Frame: Data will be made available after 1) the primary paper has been accepted for publication, or 2) the data is locked for more than 18 months, whichever comes first.
Access Criteria: De-identified scientific data generated from this study will be available to the public in the NIDA data repository, per NIDA CTN policy and the Data Management and Sharing Plan for this study.
URL: http://datashare.nida.nih.gov